CLINICAL TRIAL: NCT05990387
Title: Mirabegron and Physiological Function in Cold Environments - Aim 1
Brief Title: MIrabegron and Physiological Function in Cold Environments
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Blair D. Johnson, PhD, Associate Professor School of Public Health, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011690870; Aim 2
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Resting Energy Expenditure; Thermogenesis; Brown Adipose Tissue
MeSH Terms: interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Given once, followed by observation for up to 4 hours in a progressively cold water challenge
  Interventions: Drug: Placebo
- 100 mg Mirabegron (Experimental): Given once, followed by observation for up to 4 hours in a progressively cold water challenge
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Dose-response effect on thermogenesis
  Other Names: Myrbetriq
  Arms: 100 mg Mirabegron
Drug: Placebo — Placebo control condition
  Arms: Placebo

SUMMARY:
Many Navy diving operations are performed in cold water. Despite technical advances to improve thermal protection for cold water diving, these applications are cumbersome and do not provide complete thermal protection as thermal discomfort is subjectively reported by many Navy divers. Brown adipose tissue is highly thermogenic in humans. Therefore, activation of brown adipose tissue might improve cold water tolerance and lower thermal discomfort during cold water diving operations. Mirabegron is a beta-3-adrenergic receptor agonist that is used to treat overactive bladder. Beta-3-adrenergic receptors are located on the urinary bladder, gallbladder and brown adipose tissue. Recent evidence has demonstrated that acute mirabegron administration increases thermogenesis for ~3 hours in humans. However, it is currently not known which dose of mirabegron can increase thermogenesis for longer durations. It is also not known if mirabegron administration can improve cold water tolerance and thermal discomfort during cold water immersion. Finally, it is not known if mirabegron can increase thermogenesis during sympathetic stimulation. This project will fill these knowledge gaps by determining if acute mirabegron administration will delay the fall in core temperature and the onset of shivering during a progressive cold-water immersion challenge. This study is part of a collection of studies that will show if mirabegron is a potential ergogenic aid that can be used to improve cold water tolerance in Navy divers which will ultimately improve the likelihood of successful missions.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, cross-over experimental design. Participants will be asked to complete 3 visits to the laboratory; one informed consent/screening visit and 2 study visits. On study visit days, participants will report to the laboratory following a 12-hour fast, and 24-hour abstention from exercise, caffeine, and alcohol. During the study visits, participants will ingest either a placebo or one dose of mirabegron prior to entering our water immersion tank. Then they will be instrumented for the measurement of heart rate (3-lead ECG), blood pressure (brachial artery auscultation), core temperature (rectal thermistor), and indices of shivering (surface mechanomyography using triaxial accelerometers at 3 anatomic sites (chest, upper back, and thigh), oxygen consumption via ventilation and expired gases, and the bedside shivering assessment scale). Thermal perceptions will be assessed using Likert scales for thermal discomfort and thermal sensation. Following 10 minutes of resting baseline measurements, infrared thermography will then be used to measure skin temperature of the supraclavicular fossa as an estimate of brown adipose tissue activation and thermal perceptions will be assessed.

The measurement of supraclavicular fossa skin temperature (infrared thermography) and thermal perceptions will be assessed every 10 minutes prior to the progressive cold-water challenge. After 30 minutes of seated rest, pre-immersion measurements of heart rate, blood pressure, core temperature, shivering, and thermal perceptions will be conducted and an infrared thermography image will be taken. Then, the water immersion tank will be filled up to the participant's neck with 35 degrees C (95 degrees F) water. Heart rate, blood pressure, core temperature, and shivering indices will be continuously measured. Infrared thermography and thermal perceptions will be obtained every 5 minutes throughout the progressive cold-water challenge. The temperature of the water will be progressively lowered by ~12 degrees C every 60 minutes until the water temperature reaches 10 degrees C (50 degrees F) or until the participant can no longer tolerate the cold or if rectal temperature reaches 35.5 degrees C (95.9 degrees F). Upon completion of the progressive cold water challenge, the water in the tank will be rapidly emptied. Participants will gently towel dry and will be able to don a circulating warm water perfused suit and/or use a mylar blanket to reestablish core temperature.

Participants will be asked to return to the laboratory after 10-14 days to repeat the experiment with the drug assignment not yet received. Each participant's order of assignment to placebo or drug ingestion (prior to the cold water challenge) over the 2 study visits will be randomly assigned.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 18-40 years old
* Participate in 150 minutes or more of at least moderate intensity exercise per week during the previous 2 years

Exclusion Criteria:

* diagnosed autonomic disease
* diagnosed cardiovascular disease
* diagnosed metabolic disease
* diagnosed neurologic disease
* diagnosed endocrine disease
* diagnosed respiratory disease
* diagnosed liver dysfunction
* diagnosed kidney dysfunction
* Women who are pregnant or breastfeeding
* Individuals currently taking a medication (with the exception of birth control, including hormonal contraception) that cannot be safely discontinued for 5 biological half-lifes prior to each study visit based on consultation with the study physician.
* Current tobacco or electronic cigarette use or consistent use within the last 1 year

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blair D Johnson, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a repeated measures study design. 17 subjects provided written informed consent and were randomized. Of these subjects, 12 completed both arms of the study and 5 withdrew voluntarily (3 provided no reason for voluntarily withdrawing, 1 had a minor illness not related to the study prior to participation and chose to voluntarily withdraw, 1 voluntarily withdrew due to concerns about taking a medication).
Groups:
- Placebo First, Then Mirabegron: Placebo (two encapsulated placebo tablets) was given once followed by observation for up to 4 hours in a progressive cold water challenge. This was followed by a 10 day washout period. Then, mirabegron (two 50 mg encapsulated mirabegron tablets) was given once followed by observation for up to 4 hours in a progressive cold water challenge.
- Mirabegron First, Then Placebo: Mirabegron (two 50 mg encapsulated mirabegron tablets) was given once followed by observation for up to 4 hours in a progressive cold water challenge. This was followed by a 10 day washout period. Then, placebo (two encapsulated placebo tablets) was given once followed by observation for up to 4 hours in a progressive cold water challenge.
Period: Informed Consent/Screening Visit
Arm/Group | Placebo First, Then Mirabegron | Mirabegron First, Then Placebo
Started | 8 | 9
Completed | 5 | 7
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Period: Interventions
Arm/Group | Placebo First, Then Mirabegron | Mirabegron First, Then Placebo
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Given once, followed by observation for up to 4 hours in a progressive cold water challenge
  Placebo: Placebo control condition
  Mirabegron: 100 mg of mirabegron condition
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26 (5)

OUTCOME MEASURES:

1. Primary Outcome: Cold Temperature Deflection Point
Description: Core temperature will be continuously measured using rectal thermistors. The point at which core temperature begins to fall (i.e., deflection point) will be identified using Prism 8 software by plotting core temperature vs. water temperature.
Time Frame: Through session completion, up to 4 hours
Population: Segmental analysis was unable to identify a deflection point in 4 subjects in the placebo and 4 subjects in the 100 mg Mirabegron conditions.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Placebo | 100 mg Mirabegron
Number analyzed (Participants) | 8 | 8
degrees Celsius | 22.8 (5.67) | 22.97 (7.42)

2. Secondary Outcome: Thermogenesis - Oxygen Consumption
Description: Oxygen consumption is one measure of shivering. A pneumotach connected to a mouthpiece or facemask will be used to measure the flow of inspired and expired air. Expired gases will be sampled using oxygen and carbon dioxide sensors to determine oxygen consumption and carbon dioxide production.
Time Frame: Through session completion, up to 4 hours
Measure: Mean (Standard Deviation); unit: ml of oxygen / min / kg of body mass
Arm/Group | Placebo | 100 mg Mirabegron
Number analyzed (Participants) | 12 | 12
ml of oxygen / min / kg of body mass | 7.2 (3.1) | 7.6 (3.3)

3. Secondary Outcome: Shivering Inflection Point - Surface Mechanomyography
Description: Surface Mechanomyography is one measure of shivering. Three triaxial accelerometers adhered to the skin using adhesive tape on the chest, upper back, and thigh were used to assess shivering. The inflection point was determined using segmental analysis for each person to identify when an abrupt increase in shivering occurred.
Time Frame: Through session completion, up to 4 hours
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Placebo | 100 mg Mirabegron
Number analyzed (Participants) | 12 | 12
degrees Celsius | 24.1 (2.8) | 22.7 (3.6)

4. Secondary Outcome: Shivering Inflection Point - Bedside Shivering Scale
Description: The Bedside Shivering Scale is one measure of shivering. Two investigators will subjectively assess shivering by the participants using a Likert scale (0 = none, 3 = Severe) and the scores will be averaged. The inflection point was determined using segmental analysis for each person to identify when an abrupt increase in the bedside shivering scale occurred.
Time Frame: Through session completion, up to 4 hours
Measure: Mean (Standard Deviation); unit: degrees celsius
Arm/Group | Placebo | 100 mg Mirabegron
Number analyzed (Participants) | 12 | 12
degrees celsius | 22.1 (2.5) | 19.8 (3.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each subject after informed consent was obtained and up to their study completion (up to 6 months).
Arm/Group | Placebo | 100 mg Mirabegron
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT05990387/Prot_SAP_000.pdf